CLINICAL TRIAL: NCT05413681
Title: Metabolomic Approach During Exercise Testing in Myalgia Induced by eXercise
Acronym: Matmix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AOI 2020 RANNOU; 2020-A03296-33 (Other: 2020-A03296-33)
Record Dates: First submitted 2022-04-12; First posted 2022-06-10 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Metabolic Myopathy

STUDY DESIGN:
Intervention Model Description: Prospective study in two arms: a group of patients referred for metabolic exploration during exercise as part of their care and a group of control subjects who will perform the same explorations as the patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metabolic myopathy (Active Comparator): a supra-maximal exercise test on a cycloergometer.
  Interventions: Diagnostic Test: a supra-maximal exercise test on a cycloergometer.; Diagnostic Test: handgrip muscle activity test.
- Control : Healthy volonteers (Placebo Comparator): a supra-maximal exercise test on a cycloergometer.
  Interventions: Diagnostic Test: a supra-maximal exercise test on a cycloergometer.; Diagnostic Test: handgrip muscle activity test.

INTERVENTIONS:
Diagnostic Test: a supra-maximal exercise test on a cycloergometer. — 10 blood samples will be taken: before, during and during recovery from exercise: before the exercise test on the cycloergometer, 2 samples during exercise on the cycloergometer (middle of the threshold and peak of the exercise), 2 samples during recovery from exercise on the cycloergometer (at 2 and 10 minutes), and 1 sample at 24 hours.
Diagnostic Test: handgrip muscle activity test. — 2 bloods samples : at rest, after the 3 maximum contractions of the forearm, at 5 minute's recovery from the 30-second contraction of the grip test,

SUMMARY:
Metabolic myopathies form a group of pathologies related to a deficit of muscle energy production (enzymatic deficit) by disorder of the metabolism of carbohydrates, lipids, purines, or mitochondrial involvement related to dysfunction of complex respiratory chain. Most often, the symptomatology may include signs of "muscular" calling with cramps, contractures or exercise myalgia, more or less associated with exercise intolerance with early fatigability and rhabdomyolysis. In practice, the clinical signs are not specific and not pathognomonic, or sometimes absent with only an isolated elevation of the CPK. The diagnosis of certainty is usually based on the realization of a muscle biopsy (invasive). Unfortunately, the performance of the biopsy (definitive diagnosis of myopathy) in front of myalgia is low, hence the interest of functional explorations upstream to better specify its indication.

Given the considerable increase in muscle metabolism to physical effort, resting investigations may not uncover myo-metabolic deficit. The muscle enzymatic deficit, is therefore most often "silent" at rest and its highlighting requires to explore the patient with effort, asking him to perform an exercise test on cycloergometer and/or an isometric contraction of the forearm ('handgrip test'). Currently, only a few metabolites are dosed before and after exertion such as lactate, pyruvic acid and ammonium. Several studies in normal subjects showed the effect of physical exercise on the metabolomic signature of plasma. Our aim is to apply modern metabolomic techniques to plasma and urinary samples collected as part of the care pathway in patients referred to in the Department of Sports Medicine-Functional Explorations of the CHU in comparison with healthy volunteers).

DETAILED DESCRIPTION:
Patients will be pre-selected on the basis of their medical records and control subjects will be subjected, after signing the consent form, to a medical check-up, carried out at one of the study sites, including an interrogation on personal and family history and medication taken as well as a standard medical examination.

All subjects will be checked for compliance with the inclusion/exclusion criteria during this visit.

The subjects (patients and controls) will arrive in the morning on an empty stomach at the Sports Medicine Department of the Clermont-Ferrand University Hospital or at the Human Nutrition Unit for healthy volunteers. The subjects will be questioned about their personal and family history, about any medication they are taking, and their height and weight will be measured. The subjects will meet with a dietician to review their diet over the past 24 hours. A urine sample will be collected and divided into two aliquots: one for urinary organic acid chromatography (routine care) and one for storage for later metabolomics, transcriptomics and genomics.

Blood samples (n = 120) will be taken at the same times as during their usual care, before, during and during recovery from exercise: at rest, after the 3 maximal forearm contractions, at 1 minute of recovery from the 30-second grip-test contraction effort, before the exercise test on a cycloergometer, 2 samples during exercise on a cycloergometer (mid 'threshold' and peak of the effort), 2 samples during recovery from exercise on a cycloergometer (at 2 and 10 minutes), and 1 sample at 24 hours.

Patients will be offered to take this sample, 24 hours after the exercise test, at the Nutritional Testing Unit of the CRNH A or in their usual laboratory. If patients come to the Nutritional Testing Unit of the CRNH A for this blood test, the patients will be offered to measure their maximal muscular oxidative capacity (mVO2), using optical measurement of muscle oxygenation (near infrared spectroscopy, NIRS). If the patients do not return to the Nutritional Investigation Unit of the CRNH A for the 24-hour blood test, this measurement of maximal muscular oxidative capacity will be performed during their medical consultation to inform them of the results of their metabolic stress test (approximately 1 month later).

All the control subjects will have their blood taken at 24 hours after the exercise test at the Nutritional Investigation Unit of the CRNH A with, at the end, a measurement of their maximal muscular oxidative capacity (mVO2).

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Patient, male or female, adult or minor aged 15 years or more, referred to the Sports Medicine Department of the Clermont-Ferrand University Hospital for metabolic exploration during exercise, as part of the diagnostic work-up for one of the following clinical contexts:
* Suspicion of metabolic myopathy
* Cramps, contractures or myalgias during or after exercise
* Exercise intolerance/fatigability without obvious cause (cardiac and/or respiratory etiology in particular)
* Episode of malignant hyperthermia or rhabdomyolysis during exercise
* Unexplained elevation of CPK

For healthy subjects:

* Major subject, male or female, 18 to 50 years old.
* No chronic pathology
* No treatment (background or at the time of the examination)
* Non-smoker
* No/little alcohol consumption (<5 glasses/week), no consumption in the 48 hours before the stress test
* Non/little athletic (<2h of strenuous physical activity/week), no physical activity the day before and the day of (pre- and post-test)

For all participants:

* Able to give informed consent to participate in the research
* For minor patients, consent from the holders of parental authority
* Affiliation to the French Social Security system

Exclusion Criteria:

For healthy subjects:

* Refusal of registration in the national file of volunteers for research involving the human person.
* Subject in a period of exclusion from a previous study or having received a total amount of compensation greater than 4500 euros over the 12 months preceding the start of the trial (after verification in the File of Volunteers for Research Involving the Human Person).

For all participants:

* Contraindications to an exercise test on a cycloergometer, mainly cardiorespiratory (ATS/ACCP statement on cardiopulmonary exercise testing. Am J Respi Care Med. 2003;167:211-77.)
* Pregnant women (a pregnancy test will be performed on all participants of childbearing age on the day the exercise tests are performed) and nursing mothers.
* Refusal to sign the consent form.
* Patients under guardianship, curatorship, deprived of liberty or safeguard of justice.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Metabolomic response profile mesuring by mass spectrometer during a supra-maximal exercise test on a cycloergometer. | Before effort test
  blood samples will be taken : before the exercise test on the cycloergometer, 2 samples during exercise on the cycloergometer (middle of the threshold and peak of the exercise), 2 samples during recovery from exercise on the cycloergometer (at 2 and 10 minutes), and 1 sample at 24 hours
Metabolomic response profile mesuring by mass spectrometer during a supra-maximal exercise test on a cycloergometer. | during effort test
  blood samples will be taken : before the exercise test on the cycloergometer, 2 samples during exercise on the cycloergometer (middle of the threshold and peak of the exercise), 2 samples during recovery from exercise on the cycloergometer (at 2 and 10 minutes), and 1 sample at 24 hours
Metabolomic response profile mesuring by mass spectrometer during a supra-maximal exercise test on a cycloergometer. | 2 minutes after effort test
  blood samples will be taken : before the exercise test on the cycloergometer, 2 samples during exercise on the cycloergometer (middle of the threshold and peak of the exercise), 2 samples during recovery from exercise on the cycloergometer (at 2 and 10 minutes), and 1 sample at 24 hours
Metabolomic response profile mesuring by mass spectrometer during a supra-maximal exercise test on a cycloergometer. | 10 minutes after effort test
  blood samples will be taken : before the exercise test on the cycloergometer, 2 samples during exercise on the cycloergometer (middle of the threshold and peak of the exercise), 2 samples during recovery from exercise on the cycloergometer (at 2 and 10 minutes), and 1 sample at 24 hours
Metabolomic response profile mesuring by mass spectrometer during a supra-maximal exercise test on a cycloergometer. | 24 hours after effort test
  blood samples will be taken : before the exercise test on the cycloergometer, 2 samples during exercise on the cycloergometer (middle of the threshold and peak of the exercise), 2 samples during recovery from exercise on the cycloergometer (at 2 and 10 minutes), and 1 sample at 24 hours

SECONDARY OUTCOMES:
Metabolomic response profile mesuring by mass spectrometer to a handgrip muscle activity test. | Before grip-test
  Subjects perform a first functional test, the grip-test. This test consists of an isometric contraction of the forearm muscles. The effort is standardized by asking the subject to perform a contraction at 70% of maximum. The subject performs three maximal contractions (5 seconds) of the forearm where the catheter is inserted, spaced with 1 minute of recovery. The best value is taken as the maximum voluntary contraction force (MVCF). After 5 minutes of rest, a blood sample is taken (to ensure that the 3 maximal contractions have not modified the metabolite concentrations) and then the subject performs a 30-second contraction at 70% MVCF.
Metabolomic response profile mesuring by mass spectrometer to a handgrip muscle activity test. | 5 minutes after grip-test
  Subjects perform a first functional test, the grip-test. This test consists of an isometric contraction of the forearm muscles. The effort is standardized by asking the subject to perform a contraction at 70% of maximum. The subject performs three maximal contractions (5 seconds) of the forearm where the catheter is inserted, spaced with 1 minute of recovery. The best value is taken as the maximum voluntary contraction force (MVCF). After 5 minutes of rest, a blood sample is taken (to ensure that the 3 maximal contractions have not modified the metabolite concentrations) and then the subject performs a 30-second contraction at 70% MVCF.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice RANNOU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France